CLINICAL TRIAL: NCT00763646
Title: Phase II Study of Neoadjuvant Taxotere, Cisplatin, and 5-Fluorouracil in Patients With Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University (Other)
Responsible Party: Dr. Lorenzo Ferri, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: McG 0620; 116082
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-09

CONDITIONS: Gastric Junction Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
Keywords: Gastric or Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Docetaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Taxotere, Cisplatin, and 5-FU — Taxotere/Cisplatin/5-FU x 3 cycles (3 weeks per cycle or 9 weeks total), 1 - 2 weeks, Taxotere/Cisplatin/5-FU x 3 cycles (3 weeks per cycle or 9 weeks total)

SUMMARY:
The primary purpose of the study is to determine the impact of chemotherapy on the ability of your surgeon to completely remove the cancer as well as the impact on your survival. Furthermore the investigators will be assessing the side effects of this chemotherapy strategy. Finally the investigators will determine the ability of specialized imaging technology (PET scan) to document and predict the response of the tumor to this chemotherapy.

Standard therapy for patients with your condition usually consists of surgery (removal of the tumor) followed by combination chemotherapy and radiotherapy. More recently, standard options available to patients with cancer of the stomach or lower esophagus have been expanded to include chemotherapy without radiotherapy prior to and following surgery. While it is believed that chemotherapy prior to surgery is a good option for patients with stomach, it is not known what is the optimal chemotherapy regimen to offer patients prior to surgery to improve the likelihood of cure while limiting side-effects to patients.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of adenocarcinoma of the stomach, gastroesophageal junction (GEJ), or lower third of the esophagus.
* The tumour must be deemed by the team to be potentially resectable. This includes imaging studies (detailed below) to clinically stage the tumour and rule-out the presence of metastatic disease, and includes a preoperative laparoscopic evaluation.
* Stage IB (T1N1 only), II, IIIA, IIIB, and IV (T4N1 only)
* Life expectancy greater than 3 months
* ECOG performance status of 1 or better (i.e. restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work).
* Adequate hematologic reserve: Platelet count 100,000/L, WBC 2000/μL
* Creatinine clearance 60 ml/min, AST & ALT 2 ULN, Alkaline phosphatase 2.5 ULN, bilirubin ULN

Exclusion Criteria:

* Prior systemic therapy for gastric cancer
* Prior docetaxel-containing chemotherapy
* Pre-existing medical conditions precluding treatment, including any contraindication for major surgery
* Pregnancy or lactating mothers. Women of childbearing age must use contraception during and for 3 months following treatment.
* Unable to give informed consent
* Patients that are not able to maintain nutrition by oral consumption of food alone must have additional enteral feeding.
* Patients with macroscopic disease noted at laparoscopy
* ECOG performance status of 2 or higher
* Significant hearing impairment, as judged by the need for or use of a hearing aid. If there is any uncertainty regarding the degree of hearing impairment, an audiogram will be done. If the audiogram is grossly normal or shows only minor hearing impairment (i.e. not requiring hearing aid), the patient may be enrolled.
* Unwillingness to undergo investigations and/or treatment as outlined on the study

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-04; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To determine the impact of chemotherapy on the ability of your surgeon to completely remove the cancer as well as the impact on your survival.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Ferri, Principal Investigator — McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada